CLINICAL TRIAL: NCT01363323
Title: A Randomized, Double-Blind, Placebo/Positive Controlled, Evaluation of the Effects of MNTX on ECG Parameters and Cardiac Repolarization in Normal Volunteers
Brief Title: Effect of Methylnaltrexone (MNTX) on Electrocardiogram (ECG) Parameters and Cardiac Repolarization
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Tage Ramakrishna, M.D., Progenics Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MNTX 1106
Record Dates: First submitted 2011-05-27; First posted 2011-06-01 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — methylnaltrexone; Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arm 1 (Experimental)
  Interventions: Drug: Methylnaltrexone (MNTX)
- Arm 2 (Experimental)
  Interventions: Drug: Methylnaltrexone (MNTX)
- Arm 3 (Experimental)
  Interventions: Drug: Methylnaltrexone (MNTX)
- Arm 4 (Placebo Comparator)
  Interventions: Drug: Placebo
- Arm 5 (Active Comparator)
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Methylnaltrexone (MNTX) — Dose 1
  Arms: Arm 1
Drug: Methylnaltrexone (MNTX) — Dose 2
  Arms: Arm 2
Drug: Methylnaltrexone (MNTX) — Dose 3
  Arms: Arm 3
Drug: Placebo
  Arms: Arm 4
Drug: Moxifloxacin
  Arms: Arm 5

SUMMARY:
This study will employ a single-center, randomized, double-blind parallel-group design for MNTX and placebo, with a positive control (moxifloxacin) dosed single-blind to confirm methodology, in normal healthy male and female volunteers. Multiple ECGs will be obtained after single clinical and supratherapeutic doses of MNTX to assess ECG effects compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy and free of acute active illnesses
2. Males and females between the ages of 18 and 45 years, inclusive
3. Body mass index between 18-30, inclusive, and weight between 50-110 kgs
4. ECG within normal limits (including PR <220, QRS <110, and QTc <450 ms.)

Exclusion Criteria:

1. Previous MNTX exposure
2. Currently pregnant or nursing
3. History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological, or other medically significant disorders
4. Consumption of alcoholic beverages within 7 days prior to study confinement
5. Any evidence of congenital or familial long-QT syndrome
6. History of drug abuse of positive findings on urine drug screen
7. Known allergy or hypersensitivity to MNTX or its excipients, moxifloxacin, opioids, or related drugs or a history or relevant adverse drug reactions of any origin.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 546 (Actual)
Dates: Start 2004-11; Primary Completion 2005-01 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Effects of MNTX on QTcI duration | 3 days
  The primary objective of the study is to compare the effects of clinical and supratherapeutic doses of MNTX with the effects of placebo on QTcI duration in healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Tage Ramakrishna, MD, Study Director — Progenics Pharmaceuticals, Inc.
Locations (1):
- Progenics Pharmaceuticals, Tarrytown, New York, United States